CLINICAL TRIAL: NCT01466374
Title: A Phase IIa, Double-Blind, Randomized, Placebo-Controlled Study to Evaluate the Clinical Efficacy and Safety of Induction and Maintenance Therapy With BMS-936557 in Subjects With Active Crohn's Disease
Brief Title: Induction and Maintenance Study of BMS-936557 in Patients With Moderate to Severely Active Crohn's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IM129-008; 2011-002981-19 (EudraCT Number)
Record Dates: First submitted 2011-11-03; First posted 2011-11-08 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-09

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — BMS-936557

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Cohort 1: Induction (Experimental): Placebo
  Interventions: Drug: Placebo
- Cohort 2: Induction (Experimental): Anti-IP-10 Antibody
  Interventions: Drug: BMS-936557 (Anti-IP-10 Antibody)
- Cohort 3: Induction (Experimental): Anti-IP-10 Antibody
  Interventions: Drug: BMS-936557 (Anti-IP-10 Antibody)
- Cohort 1: Maintenance (Experimental): Placebo
  Interventions: Drug: Placebo
- Cohort 2: Maintenance (Experimental): Anti-IP-10 Antibody
  Interventions: Drug: BMS-936557 (Anti-IP-10 Antibody)
- Cohort 3: Maintenance (Experimental): Anti-IP-10 Antibody
  Interventions: Drug: BMS-936557 (Anti-IP-10 Antibody)
- Cohort 1: Open Label (Experimental): Anti-IP-10 Antibody
  Interventions: Drug: BMS-936557 (Anti-IP-10 Antibody)

INTERVENTIONS:
Drug: Placebo — Normal Saline, Intravenous (IV), 0 mg, Once a week for the first week and every other week thereafter, 11 weeks
  Arms: Cohort 1: Induction
Drug: Placebo — Normal Saline, Intravenous, 0 mg, Every other week, Up to 337days
  Arms: Cohort 1: Maintenance
Drug: BMS-936557 (Anti-IP-10 Antibody) — Solution for IV administration, Intravenous, 10 mg/kg, Once a week for the first week and every other week thereafter, 11 weeks
  Other Names: Anti-IP-10 Antibody
  Arms: Cohort 2: Induction
Drug: BMS-936557 (Anti-IP-10 Antibody) — Solution for IV administration, Intravenous, 20 mg/kg, Once a week for the first week and every other week thereafter, 11 weeks
  Other Names: Anti-IP-10 Antibody
  Arms: Cohort 3: Induction
Drug: BMS-936557 (Anti-IP-10 Antibody) — Solution for IV administration, Intravenous, 7.5 mg/kg, Every other week, Up to 337 days
  Arms: Cohort 2: Maintenance
Drug: BMS-936557 (Anti-IP-10 Antibody) — Solution for IV administration, Intravenous, 15 mg/kg, Every other week, Up to 337 days
  Arms: Cohort 3: Maintenance
Drug: BMS-936557 (Anti-IP-10 Antibody) — Solution for IV administration, Intravenous, 15 mg/kg or optimal dose, Every other week, Open
  Arms: Cohort 1: Open Label

SUMMARY:
The purpose of this study is to determine whether BMS-936557 is effective for the treatment of moderate to severely active Crohn's Disease in patients who have had insufficient response and/or intolerance to conventional therapy for Crohn's Disease.

DETAILED DESCRIPTION:
Anti-IP10: Anti Interferon-inducible ligand 10

ELIGIBILITY:
Inclusion Criteria:

* Adults subjects with confirmed Crohn's Disease (CD) for at least 3 months
* Moderate to severely active CD as defined by Crohn's Disease Activity Index (CDAI) 220 to 450
* In the past have had insufficient response and or intolerance to ≥ 1 of the conventional therapy (immunosuppressants, corticosteroids and/or approved biologic therapy)

Exclusion Criteria:

* Ulcerative colitis (UC) or indeterminate colitis
* Short bowel syndrome
* Known stricture or noninflammatory stenosis leading to symptoms of obstruction
* Current stoma or current need for colostomy or ileostomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2011-12; Primary Completion 2014-06 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Clinical remission (CDAI score of <150) | Week 11
  CDAI: Crohn's Disease Activity Index

SECONDARY OUTCOMES:
Proportion of subjects in clinical remission (defined by an absolute CDAI score < 150) | Week 7 and Week 11
Proportion of subjects in clinical response (defined as CDAI score reduction from Baseline of ≥ 100 points or an absolute CDAI score of < 150) | Week 7 and Week 11
Mean change from baseline in Inflammatory Bowel Disease Questionnaire (IBDQ) | Week 11
Safety of BMS-936557 in the induction period defined by proportion of subjects reporting AE, SAEs, AEs leading to discontinuation, and markedly abnormal laboratory values | Week 11
  AE - Adverse Event SAE - Serious Adverse Event

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (30):
- United States (10):
  - Southern California Medical Gastroenterology Group, Santa Monica, California
  - Shafran Gasteroenterology Center, Winter Park, Florida
  - Gastroenterology Research Of New Orleans, Hammond, Louisiana
  - Metropolitan Gastroenterology Group, Pc, Chevy Chase Cr, Chevy Chase, Maryland
  - Midwest Center For Clinical Research, Lees Summit, Missouri
  - Nyu Langone Long Island Clinical Research Associates, Great Neck, New York
  - Mount Sinai School Of Medicine, New York, New York
  - University Of North Carolina At Chapel Hill, Chapel Hill, North Carolina
  - Consultants For Clinical Research, Cincinnati, Ohio
  - Gastroenterology Research Of San Antonio, San Antonio, Texas
- Belgium (2):
  - Local Institution, Brussels
  - Local Institution, Leuven
- France (6):
  - Local Institution, Amiens
  - Local Institution, Clichy
  - Local Institution, Nice
  - Local Institution, Pessac
  - Local Institution, Rouen
  - Local Institution, Vandœuvre-lès-Nancy
- Hungary (2):
  - Local Institution, Budapest
  - Local Institution, Debrecen
- Israel (3):
  - Local Institution, Haifa
  - Local Institution, Kfar Saba
  - Local Institution, Nazareth
- Poland (3):
  - Local Institution, Krakow
  - Local Institution, Rzeszów
  - Local Institution, Warsaw
- University Of Puerto Rico School Of Medicine, San Juan, Puerto Rico
- South Africa (3):
  - Local Institution, Overport, KwaZulu-Natal
  - Local Institution, Claremont, Western Cape
  - Local Institution, Panorama, Western Cape

REFERENCES:
- [Derived] Sandborn WJ, Rutgeerts P, Colombel JF, Ghosh S, Petryka R, Sands BE, Mitra P, Luo A. Eldelumab [anti-interferon-gamma-inducible protein-10 antibody] Induction Therapy for Active Crohn's Disease: a Randomised, Double-blind, Placebo-controlled Phase IIa Study. J Crohns Colitis. 2017 Jul 1;11(7):811-819. doi: 10.1093/ecco-jcc/jjx005. PMID 28333187
- [Derived] Khanna R, Zou G, D'Haens G, Rutgeerts P, McDonald JW, Daperno M, Feagan BG, Sandborn WJ, Dubcenco E, Stitt L, Vandervoort MK, Donner A, Luo A, Levesque BG. Reliability among central readers in the evaluation of endoscopic findings from patients with Crohn's disease. Gut. 2016 Jul;65(7):1119-25. doi: 10.1136/gutjnl-2014-308973. Epub 2015 May 2. PMID 25935574
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx